CLINICAL TRIAL: NCT06558474
Title: Optimization of Percutaneous Coronary Intervention After Stent Implantation With Liberal Use of High-pressure Non-compliant Balloon Post-dilatation Versus Contemporary Practice
Brief Title: Optimization of Percutaenous Coronary Intervention With Liberal Use of Post-dilatation
Acronym: OPTIMIZE-PCI
Status: Recruiting | Type: Observational
Sponsor: Cathreine BV (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Koen Teeuwen, Principal investigator, Cathreine BV
Other Study IDs: CathreineBV
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; coronary artery disease; stent optimization; post-dilatation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-intervention/implementation cohort: In the first phase, data additional to the national PCI registry will be analyzed retrospectively from all patients receiving PCI from January 2021 to January 2022. Data on the percentage of use of post-dilatation using high-pressure non-compliant (HPNC) balloon by the individual interventional cardiologist will be collected. This will establish a benchmark from which individual interventional cardiologists must increase their use of post-dilatation.
- Post-intervention/implementation cohort: During this implementation phase, all individual PCI operators of the participating centres will be informed to liberally use post-dilatation for stent optimization during PCI. Operators are requested to increase their use of post-dilatation with at least 20% or use post-diltation in at least 85% of the PCI's. Throughout the project, individual participating operators will receive individual feedback on the percentage use of post-dilatation with prospective data collection after 2, 4, 6, 9 and 12 months. Based on this result, the implementation process will be refined as necessary. The duration of this phase will be approximately 1 year per centre.
  Eventually a retrospective observational anlaysis, comparing the two cohorts, will be conducted to evaluate whether adopting this strategy has led to improved clinical outcomes after PCI in terms of major adverse cardiac events.
  Interventions: Behavioral: Liberal post-dilatation strategy during PCI

INTERVENTIONS:
Behavioral: Liberal post-dilatation strategy during PCI — A liberal post-dilatation strategy for stent optimization during PCI will be implemented in multiple centers in the Netherlands.
  This include an increase of post-dilatation use of at least 20% per operator, or a percentage of post-dilatation of at least 85%.
  Operators will be asked to enforce a very low threshold for post-dilatation in general, with a mandatory HPNC post-dilatation for the following indications:
  * In case of any calcification
  * Delta of ≥ 0.5mm between the distal and proximal reference diameter of the treated coronary segment
  * Stent length >24 mm
  * Signs of incomplete stentframe-deployment on angiography or StentBoost
  * In case of CTO
  * In case of bifurcation PCI (Left main and non-left main)
    * Proximal Optimisation Technique (POT) with NC balloon
    * Final Kissing Balloon dilatation (FKB) with preferentially first sequential high-pressure inflations and final low pressure kiss both with NC balloons
  Groups: Post-intervention/implementation cohort

SUMMARY:
To achieve optimal long-term clinical results after percutaneous coronary intervention (PCI), adequate deployment of stents is essential. Thorough expansion of the stent and full apposition of stent struts against the vessel wall are determining factors for preventing stent thrombosis and restenosis for bare-metal as well as drug-eluting stents (DES). Standard coronary angiography is limited in assessing accurate vessel size and characterizing tissues and calcium load. Therefore, stent underexpansion frequently occurs after stent deployment.

Post-dilation is often performed to achieve optimal stent expansion and reduce stent malapposition of stent struts, aiming to reduce stent thrombosis and restenosis both short term as long term. However, there are limited studies that have explored the effect of post-dilatation for stent optimization on clinical outcomes. As a result of the restricted evidence, there is no consensus whether post-dilatation should be used routinely in clinical practice and the extent to which post-dilatation is being utilized remains unclear.

For this reason, the OPTIMIZE PCI was designed, a national registry-based quality improvement project to implement a liberal post-dilatation strategy in multiple PCI centers in the Netherlands. As part of the OPTIMIZE-PCI, a retrospective observational analysis will eventually be conducted to evaluate whether adopting this strategy has led to improved clinical outcomes after PCI in terms of major adverse cardiac events.

DETAILED DESCRIPTION:
The Netherlands Heart Registration (NHR) is an independent organization in which Dutch hospitals prospectively register standard sets of baseline, procedural and outcome data for all invasive cardiac procedures, including PCI. Data provided to the NHR are extensively checked on completeness and quality, reviewed with audit reports by independent trained research nurses and discussed by cardiologists in registration committees. Multiple audits are conducted annually by the NHR for data validation and verification. A waiver for informed consent for analysis with the data of the NHR data registry is obtained.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old who undergo PCI for any indication are included in the register of the Netherlands Heart Registration and therefore included in the final analysis of this project

Exclusion Criteria:

- If a patient has multiple PCIs within 365 days, only the first procedure is included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population exists of patients registered in our national PCI registration of the Netherlands Heart Registration after receiving PCI. All indications are included (ACS and non-ACS, OHCA, cardiogenic shock), resulting in an all-comer population
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of target vessel revascularization, myocardial infarction and all-cause mortality | 30 day
  The primary composite end point of major adverse cardiac events is the occurrence of target vessel revascularization, myocardial infarction and all-cause mortality.

SECONDARY OUTCOMES:
All cause mortality | 30 days, 1 year
  all cause mortality, confirmed by verifying the vital status of a patient in the Personal Records Database.
Target vessel revascularization | 30 days and 1 year
  Target vessel revascularization, defined as a revascularization by percutaneous coronary intervention or coronary artery bypass grafting in the same vessel(s) that had been treated at the index procedure, excluding staged procedures.
Myocardial infarction | 30 day
  Myocardial infarction, defined as an increase and/or decrease in one or more cardiac biomarkers by at least one value above the 99th percentile of the upper limit where at least one of the following symptoms is present: 1) symptoms appropriate to ischemia, 2) new significant ST-segment or T-wave abnormalities or bundle branch block, 3) development of pathological Q-waves on the electrocardiogram (ECG), 4) imaging demonstrated new loss of viable myocardial tissue or new wall motion abnormalities, 5) identification of intracoronary thrombus on angiography or autopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] van Beek KAJ, Timmermans MJC, Derks L, Cheng JM, Kraaijeveld AO, Arkenbout EK, Schotborgh CE, Brouwer J, Claessen BE, Lipsic E, Polad J, van Nunen LX, Sjauw K, van Veghel D, Tonino PA, Teeuwen K; 'on behalf of the PCI registration committee of The Netherlands Heart Registration'. Contemporary Use of Post-Dilatation for Stent Optimization During Percutaneous Coronary Intervention; Results From the Netherlands Heart Registration. Catheter Cardiovasc Interv. 2025 Mar;105(4):870-877. doi: 10.1002/ccd.31404. Epub 2025 Jan 8. PMID 39777867
- [Background] Slingerland SR, van Beek KAJ, Schulz DN, van Steenbergen GJ, Brouwer T, Stoel M, Vlaar PJ, Tonino PA, Dekker L, van Nunen LX, Teeuwen K, van Veghel D. Results of systematic patient outcome monitoring: Does post-dilatation during angiography-guided percutaneous coronary intervention improve clinical outcomes? Hellenic J Cardiol. 2025 Mar-Apr;82:26-33. doi: 10.1016/j.hjc.2023.11.004. Epub 2023 Nov 16. PMID 37979617